CLINICAL TRIAL: NCT07225543
Title: Scavenging IsoLGs in Autoimmune Disease: a Proof-of-concept Clinical Study
Brief Title: 2-HOBA in Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michelle Ormseth, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 250944; 1P01HL174442-01A1 (NIH)
Record Dates: First submitted 2025-11-04; First posted 2025-11-06 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Systemic Lupus Erthematosus (SLE)
Keywords: systemic lupus erythematosus; SLE; lupus; oxidative stress; hypertension; blood pressure; NETosis; isolevuglandins
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Hypertension | interventions — 2-(aminomethyl)phenol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo First (Experimental): Placebo for first 4 weeks, then washout for 4 weeks, and then 2-HOBA acetate for 4 weeks
  Interventions: Drug: 2-HOBA acetate (2-Hydroxybenzlamine acetate); Drug: Placebo
- 2-HOBA First (Experimental): 2-HOBA acetate for first 4 weeks, then washout for 4 weeks, and then placebo for 4 weeks
  Interventions: Drug: 2-HOBA acetate (2-Hydroxybenzlamine acetate); Drug: Placebo

INTERVENTIONS:
Drug: 2-HOBA acetate (2-Hydroxybenzlamine acetate) — 2-HOBA acetate (2-Hydroxybenzlamine acetate) 750mg (provided as three 250mg capsules) three times per day
  Other Names: 2-hydroxybenzylamine; 2-HOBA; salicylamine; IUPAC name: 2-(aminomethyl)phenol
Drug: Placebo — Placebo (provided as three capsules) three times per day
  Other Names: indentical placebo

SUMMARY:
This is a phase II randomized, placebo-controlled, double-blind, cross-over study to determine the effect of isolevuglandin (IsoLG) scavenging by 2-HOBA on blood pressure and immune activation in patients with SLE. 42 patients with stable SLE will be randomized to treatment sequence to receive placebo or 750mg 2-HOBA three times a day for 4 weeks followed by a 4 week washout and then 4 weeks of the other agent.

Primary outcome measures include change in 24-hour blood pressure and NETosis. This study will provide mechanistic information on the role of IsoLGs in autoimmune disease-associated hypertension and immune activation.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an inflammatory autoimmune disease with a markedly increased prevalence of not only hypertension but also resistant hypertension. Hypertension, along with other factors, leads to a 2 to 3-fold increase in risk of cardiovascular disease in SLE. Other than glucocorticoids and immunosuppression, there are few therapeutic options for patients with SLE and none that are known to have a beneficial effect on hypertension and cardiovascular disease; in fact, glucocorticoids have substantial deleterious effects. The increased prevalence of hypertension and its greater severity in SLE patients are unexplained; however, work from our group and others increasingly implicates activation of the immune system in the pathogenesis of hypertension. Moreover, our data suggest that downstream products of oxidative stress, specifically isolevuglandins (IsoLGs), drive immune activation and hypertension.

IsoLGs are highly reactive dicarbonyl products of oxidative stress that bind covalently to proteins causing conformational changes rendering them immunogenic and proinflammatory. Two decades of work at Vanderbilt led to the identification of 2-hydroxybenzylamine (2-HOBA) as a highly effective scavenger of reactive dicarbonyls such as IsoLGs. Scavenging reactive dicarbonyls is preferable to using antioxidants because reactive oxygen species are necessary for normal cellular function. In animal models of SLE, hypertension, and atherosclerosis 2-HOBA reduced inflammation, neutrophil extracellular traps (NETosis), blood pressure, and atherosclerosis, and in human phase I clinical studies with healthy volunteers it was well tolerated.

This is a mechanistic, proof-of-concept phase II study with a randomized, placebo-controlled, double-blind, cross-over design to determine the effect of IsoLG scavenging by 2-HOBA on blood pressure and immune activation in patients with SLE. 42 patients with stable SLE will be randomized to treatment sequence to receive placebo or 750mg 2-HOBA three times a day for 4 weeks followed by a 4 week washout and then 4 weeks of the other agent. Comparing 2-HOBA and placebo arms, primary outcomes include change in 24-hour blood pressure and immune activation measured by NETosis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 years
* Meeting the 2019 European League Against Rheumatism/ American College of Rheumatology classification criteria for SLE32
* No change in immunosuppressants ≥3 months
* Stable prednisone (or equivalent) dose ≤ 20mg/ day for ≥ 1 month
* Elevated blood pressure defined as >120 and < or = 160 mmHg systolic or >80 and < or = 110 mmHg diastolic blood pressure at screening visit
* No change in anti-hypertensive dose ≥2 weeks
* Willingness to stop NSAIDs for ≥2 weeks before and throughout the study
* If of childbearing potential, willingness to use effective birth control throughout the study and 4 weeks after completion of the study (examples: condom, diaphragm, oral contraceptive pill, intrauterine device)

Exclusion Criteria:

* Pregnant or breastfeeding
* Active cancer except for non-melanoma skin cancer
* Prior diagnosis of liver cirrhosis or the following abnormal liver function studies: AST or ALT >1.5x the upper limit of normal or total bilirubin ≥1.5 mg/dl
* Active infection requiring medical intervention
* Major surgery in ≤ 3 months
* Aspirin allergy
* Use of MAO-I
* Estimated creatinine clearance <30 ml/min
* Known atrial fibrillation
* Severe comorbid condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
24-hour systolic blood pressure | Measured at the beginning and end of each phase at weeks 0, 4, 8, and 12.
  Investigators will measure change in 24-hour systolic blood pressure
NETosis | Measured at beginning and end of each phase at weeks 0, 4, 8, and 12.
  Investigators will measure change in NETosis by ELISA assessing circulating NET concentration

CONTACTS AND LOCATIONS:
Overall Officials: Michelle J Ormseth, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The following data files will be produced:
  * Demographic/ clinical data such as age, race, sex, SLE disease activity measures, and medication use
  * Standard clinical laboratory measurements such as complete blood count, complete metabolic panel, complement C3 and C4, dsDNA antibody titer, erythrocyte sedimentation rate, urinalysis, spot urine protein and creatinine.
  * 24-hour blood pressure measurements
  * NETosis data
  * type 1 interferon signature Identifiable data will be de-identified and anonymized prior to sharing. Given the rarity of the disease, small geographic area of recruitment, and very specific manifestations of SLE in individual patients, the risk of re-identification of participants is real. Thus, to ensure privacy concordant with the requirements of the institutional review board, information on specific SLE manifestations will not be shared and demographic variables with few participants may be collapsed/ aggregated (e.g. age, race) to anonymize data.
Supporting Information: Study Protocol
Time Frame: Data will be made available upon publication of study results or end of the performance period, whichever comes first. The data shared will be archived and available on the Vivli platform for request by researchers for a minimum of 10 years after contribution.
Access Criteria: The Vivli platform has multiple levels of protection for managing human participant data. Each user must sign a Data Use Agreement and there is an established policy for managing violations.